CLINICAL TRIAL: NCT03337633
Title: Effects of Menu Design on Psychophysiological Measures of Cognitive Load and Food Ordering Outcomes
Brief Title: Effects of Restaurant Menu Design on Food Ordering Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Kathryn Kaiser, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: X140313004
Record Dates: First submitted 2017-10-18; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Food Preferences
Keywords: cognitive load; galvanic skin response; meal size; kilocalories; menu design
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Parallel arm randomized controlled trial
Who Masked: Participant
Masking Description: Participants were blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment 1 Easy (Active Comparator): For the first experiment, subjects in this arm received the "easy" menu during the protocol.
  Interventions: Behavioral: Menu design
- Experiment 1 Hard (Active Comparator): For the first experiment, subjects in this arm received the "hard" menu during the protocol.
  Interventions: Behavioral: Menu design
- Experiment 2 Easy (Active Comparator): For the second experiment, subjects in this arm, who qualified as restrained eaters and were asked to fast for 8 hours overnight, received the "easy" menu during the protocol.
  Interventions: Behavioral: Menu design
- Experiment 2 Hard (Active Comparator): For the second experiment, subjects in this arm, who qualified as restrained eaters and were asked to fast for 8 hours overnight, received the "hard" menu during the protocol.
  Interventions: Behavioral: Menu design

INTERVENTIONS:
Behavioral: Menu design — Participants were given 5 minutes to order a hypothetical meal from the assigned test menu by circling all items they wanted to order.

SUMMARY:
High cognitive load activities can influence energy intake from food. It is unknown how restaurant menu designs may affect patrons in terms of cognitive demand and subsequent ordering of food.Objective: Our objective was to develop and experimentally test menu designs that differ in cognitive load to test the subjective and objective stress measures on food ordering.

DETAILED DESCRIPTION:
For the first experiment, a parallel randomized trial of healthy young adults (n= 30) was conducted to compare ordering from one of two menu designs (easy - E, hard - H) developed in a prior pilot study. In the second experiment, restrained eaters were specifically recruited and asked to fast before the experiment to determine the influence of cognitive load of menus on energy ordered (n=31). Galvanic skin response was used as an objective proxy for relative cognitive load, and questionnaires were used to assess perceptions of the menus. The main outcomes were the number of items ordered and total energy of the items ordered (in kilocalories).

ELIGIBILITY:
Experiment 1

Inclusion Criteria:

* Normal vision or corrective lenses
* Normal hearing or a hearing aid
* A moderate level of English proficiency or greater
* Free from current food restrictions

Exclusion Criteria:

* Unwilling/uninterested in participation
* Currently taking any β-blocker medications
* Any serious skin conditions on the hands (because of galvanic skin sensors worn for the protocol)

Experiment 2

Inclusion Criteria:

* Normal vision or corrective lenses
* Normal hearing or a hearing aid
* A moderate level of English proficiency or greater
* Free from current food restrictions
* Qualifying as a restrained eater by the Cognitive Restraint scale on the Eating Inventory (score of 6 for men and 10 for women)

Exclusion Criteria:

* Unwilling/uninterested in participation
* Currently taking any β-blocker medications
* Any serious skin conditions on the hands (because of galvanic skin sensors worn for the protocol)

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Total Number of Items Ordered | During the 5-minute menu ordering task
  Total number of items ordered off assigned menu
Total Energy of Items ordered | During the 5-minute menu ordering task
  Total Energy (kcals) of items ordered off assigned menu

SECONDARY OUTCOMES:
Subjective ratings of difficulty of using assigned menu to order a meal | Immediately (1 minute) following the 5-minute menu ordering period
  Assessed by NASA Task Load Index questionnaire
Galvanic Skin Response | During the 5-minute menu ordering task
  An objective proxy for relative cognitive load; this measure has been shown to be positively correlated with psychological stress or cognitive challenge as mediated by sympathetic nervous system activity

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Kaiser, PhD, Principal Investigator — University of Alabama at Birmingham, Asst. Professor, Dept of Health Behavior

IPD SHARING:
Plan to Share IPD: Yes
Pending approval by the University of Alabama at Birmingham's Institutional Review Board (IRB), which we have received for other studies and anticipate receiving here, we will prepare transportable de-identified raw databases and codebooks, which will contain the raw data used in any paper we publish from the proposed research. We will publically deposit such raw data for access by others without restriction in a public repository such as ICPSR. For any investigator requesting data we have not yet published, we will be glad to provide de-identified data and codebooks to the investigators provided that the proposed use does not conflict with our intentions for use.
Supporting Information: ICF, Analytic Code
Time Frame: Materials will be posted after publication of study results.
Access Criteria: Data and supporting materials will be freely available to anyone with access to openICPSR.